CLINICAL TRIAL: NCT06559020
Title: Predictors for Opting for Kangaroo Mother Care in Pakistan and Infant Development Outcomes Based on a Quasi-Experimental Intervention
Brief Title: Predictors and Outcomes of Kangaroo Mother Care: A Quasi-Experimental Study in Pakistan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Services Institute of Medical Sciences, Pakistan (Other Government)
Responsible Party: Principal Investigator, Tayyiba Wasim, Professor Obstetrics & Gynaecology, Services Institute of Medical Sciences, Pakistan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB/2023/1099/SIMS
Record Dates: First submitted 2024-08-13; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Low Birth Weight Infants; Preterm Infants
Keywords: Kangroo mother care; Infant development; Breast feeding; Neonatal death; Vaccination; Pakistan
MeSH Terms: conditions — Breast Feeding; Perinatal Death

STUDY DESIGN:
Intervention Model Description: This study employs a quasi-experimental design with parallel assignment. Participants were self-selected into two groups: one receiving Kangaroo Mother Care (KMC) and the other receiving Conventional Care (CC). The intervention was applied without randomization, and both groups were followed for one year to assess differences in growth, developmental milestones, breastfeeding practices, vaccination status, and mortality among low birth weight and preterm infants.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- kangroo mother care (Experimental): he KMC group will receive continuous skin-to-skin contact between mother and infant for 24 hours a day, with support and training in kangaroo positioning and exclusive breastfeeding.
  Interventions: Behavioral: Kangroo mother care
- conventional care (No Intervention): The control group will receive conventional neonatal care, which includes placing newborns in open cots with appropriate heating or cooling based on weather conditions. Mothers will receive guidance on the benefits of exclusive breastfeeding and support to initiate breastfeeding, but will not have the structured kangaroo mother care provided to the experimental group.

INTERVENTIONS:
Behavioral: Kangroo mother care — Kangaroo Mother Care (KMC) involves continuous skin-to-skin contact between the mother (or another family member) and the infant, aimed at promoting thermal regulation, breastfeeding, and bonding. In this study, KMC was initiated in the hospital and continued at home for a minimum of 8 hours daily.
  Arms: kangroo mother care

SUMMARY:
This quasi-experimental study evaluated the impact of Kangaroo Mother Care (KMC) versus Conventional Care (CC) on the growth, developmental milestones, breastfeeding, vaccination, and mortality of low birth weight infants in Services Hospital Lahore, Pakistan. A total of 400 infants were enrolled and followed for one year.

DETAILED DESCRIPTION:
This quasi-experimental study was conducted in the Obstetrics and Gynecology Department of Services Institute of Medical Sciences (SIMS), Lahore, Pakistan, to compare the impact of Kangaroo Mother Care (KMC) versus Conventional Care (CC) on low birth weight infants. A total of 400 infants (200 in each group) born between January 2020 and December 2022 were included in the study, with participants selected based on specific inclusion criteria and informed consent obtained. KMC involved continuous skin-to-skin contact between mother and infant during the hospital stay and continued at home for at least 8 hours daily. The follow-up schedule included appointments at six weeks after birth, monthly visits until six months of age, and quarterly visits until the infants reached one year of age. During these visits, the study collected data on infant growth, developmental milestones, breastfeeding practices, and vaccination status. The study was ethically approved by the research ethics committee, and data collection was conducted during scheduled follow-up visits to the outpatient department.

ELIGIBILITY:
Inclusion Criteria:

* women who were able to follow the program instructions,
* permanent residents of Lahore and its periphery and willing to be part of program for the one-year time period,
* live newborn babies delivered either vaginally or through caesarean section with birth weight of 1.5 to 2 kg,
* gestational age between 28 to 36 weeks.

Exclusion Criteria:

* an infant or mother diagnosed with a life-threatening ailment, major disease, or major malformations,
* early-detected major conditions arising from perinatal problems, such as severe hypoxic-ischemic encephalopathy, pulmonary hypertension,
* incidence of severe infection measured as nosocomial infections requiring systemic antibiotics or infections, severe respiratory distress, and hypothermia episodes (temperature less than 35C).

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Duration of Breastfeeding | from 2 hours to 1 year
  breastfeeding initiation within 2 hours, exclusive breastfeeding for 6 months, breastfeeding up to one year
Number of babies with complete vaccination | 1 year
  infant receiving all scheduled vaccinations within their first year of life
Average weight of baby | 1 year
  Weight of infant in Kg at birth, 6 weeks, 1 year, 6 months, and 1 year
average length of infant | 1 year
  Length of infant in cms at birth, 6 weeks, 1 year, 6 months, and 1 year
Average head circumference of infant | 1 year
  Head circumference of infant in cms at birth, 6 weeks, 1 year, 6 months, and 1 year
Number of babies Holding head up | 3 months
  baby able to hold their head up
Number of babies Sitting without support | 6 months
  Baby gets into sitting position without help
Number of babies roll over | 8 months
  baby able to roll from side to side
Number of babies crawling | 10 months
  baby able to move forward on hands and knees
Number of babies babbles | 6 months
  baby able to produce repititive incomprehensible sounds
Number of babies produce 2 syllable sounds | 9 months
  baby able to produce words that have two definite sounds
cumulative Mortality rate | 1 year
  Death of baby

SECONDARY OUTCOMES:
Number of babies with Hypothermia | 72 hours
  core body temperature less than 35 degree celsius
Number of babies with Sepsis | 72 hours
  infection leading to life threatening inflammatory response

CONTACTS AND LOCATIONS:
Overall Officials: Tayyiba Wasim, FCPS, Principal Investigator — Services Institute of Medical Sciences, Pakistan
Locations (1):
- Services Institute of Medical sciences, Lahore, Punjab Province, Pakistan